CLINICAL TRIAL: NCT03317301
Title: a Multicenter, Randomized, Double-blinded, Active-controlled, Parallel, Phase Ⅲ Study to Evaluate the Efficacy and Safety of HL151 Versus Talion Tab. in Pruritus Cutaneus
Brief Title: Evaluate the Efficacy and Safety of HL151 Versus Talion Tab. in Pruritus Cutaneus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL_HL151_302
Record Dates: First submitted 2017-10-12; First posted 2017-10-23 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2017-10

CONDITIONS: Pruritus
Keywords: Pruritus cutaneus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental: 2 times a day(Day, Night), 2 weeks of treatment / Day: HL151 (1Tab)+Talion Tab (Placebo)(1Tab), Night: HL151 (Placebo)(1Tab)+Talion Tab (Placebo)(1Tab)
  Interventions: Drug: HL151
- Active comparator (Active Comparator): Comparator: 2 times a day(Day, Night), 2 weeks of treatment / Day: HL151 (Placebo)(1Tab)+Talion Tab (1Tab), Night: HL151 (Placebo)(1Tab)+Talion Tab (1Tab)
  Interventions: Drug: Talion Tab

INTERVENTIONS:
Drug: HL151 — 2 times a day(Day, Night), 2 weeks of treatment / Day: HL151 (1Tab)+Talion Tab (Placebo)(1Tab), Night: HL151 (Placebo)(1Tab)+Talion Tab (Placebo)(1Tab)
  Arms: Experimental
Drug: Talion Tab — 2 times a day(Day, Night), 2 weeks of treatment / Day: HL151 (Placebo)(1Tab)+Talion Tab (1Tab), Night: HL151 (Placebo)(1Tab)+Talion Tab (1Tab)
  Arms: Active comparator

SUMMARY:
a Multicenter, Randomized, Double-blinded, Active-controlled, Parallel, Phase Ⅲ Study to Evaluate the Efficacy and Safety of HL151 versus Talion Tab. in Pruritus cutaneus.

- Endpoint: VAS Score Change, Investigator's assessment of overall treatment

ELIGIBILITY:
Inclusion Criteria:

1. Both gender, 19 years ≤ age
2. Patients with pruritus due to the following diseases

   ① acute eczema, chronic eczema, monetary eczema, sebaceous deficiency eczema

   ② contact dermatitis, atopic dermatitis, seborrheic dermatitis, neurodermatitis

   ③ Acute prurigo (Strofus, Urticaria, lichen urticatus), subacute prurigo, chronic prurigo (nodular prurigo)

   ④ systemic skin pruritus, focal skin pruritus
3. In visit 2, during the run-in period previous week the VAS score of day and night time were 2 or more average points per day (maximum 4 points)
4. Those who can ability to record subject diary
5. Written consent voluntarily to participate in this clinical trial after understanding and detailed explanation about this clinical trial

Exclusion Criteria:

1. Patients with pruritus due other medical causes (liver disease, heart failure, etc.)
2. Among patients with skin disease, malignant tumors and patients with chronic urticaria skin disease
3. Patients with systemic infection symptoms at the time of clinical trials
4. Asthmatic patients requiring steroid treatment
5. Patients with Spastic diseases such as epilepsy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in VAS(Visual Analogue Scale) score at 2nd week after clinical drug administration compared to baseline | Visit 2 (0 week), Visit 3 (1 week), Visit 4 (2 weeks)
  VAS score: 0 Point ~ 10 Point (asymptomatic ~ Maximum pruritus) Evaluation period: Visit 2 (0 week), Visit 3 (1 week), Visit 4 (2 weeks)

SECONDARY OUTCOMES:
Changes in VAS(Visual Analogue Scale) score at 1st week after clinical drug administration | Visit 2 (0 week), Visit 3 (1 week)
  VAS score: 0 Point ~ 10 Point (asymptomatic ~ Maximum pruritus)
  * Evaluation period: Visit 2 (0 week), Visit 3 (1 week)
Changes in VAS(Visual Analogue Scale) score at 1st and 2nd week(Day) after clinical drug administration compared to baseline | Visit 2 (0 week), Visit 3 (1 week), Visit 4 (2 weeks
  VAS score: 0 Point ~ 10 Point (asymptomatic ~ Maximum pruritus)
  * Evaluation period: Visit 2 (0 week), Visit 3 (1 week), Visit 4 (2 weeks
Changes in VAS(Visual Analogue Scale) score at 1st and 2nd week after clinical drug administration compared to baseline | Visit 2 (0 week), Visit 3 (1 week), Visit 4 (2 weeks)
  VAS score: 0 Point ~ 10 Point (asymptomatic ~ Maximum pruritus)
  * Evaluation period: Visit 2 (0 week), Visit 3 (1 week), Visit 4 (2 weeks)
Investigator's assessment of overall treatment(Cochran-Mantel-Haenszel method) | Visit 4 (2 weeks)
  VAS score: 0 Point ~ 10 Point (asymptomatic ~ Maximum pruritus)
  * Evaluation period: Visit 4 (2 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang Univ. Guri Hospital, Guri-si, Kyeonggi-do, South Korea